CLINICAL TRIAL: NCT02794779
Title: Minimum Oxytocin Dose for Cesarean During Labor: Adaptative Clinical Trial
Acronym: MODCL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, MD, MSc, Brasilia University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: anestesiatccthiago1416
Record Dates: First submitted 2016-06-04; First posted 2016-06-09 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Cesarean Section During Labor
Keywords: cesarean section; labor; oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rule of three (Experimental): Intravenous bolus infusion of oxytocin 3UI followed by re-asessment of uterine tone by obstetrician after 3 minutes. Infusion stops when uterine tone is adequate and is repeated if inadequate to the maximum of 9UI (3 bolus infusions). If uretine tone is inadequate after 9UI then other methods for preventing bleeding will be used.
  Interventions: Drug: Oxytocin
- Continuous infusion (Active Comparator): Continuous infusion of variable rate if 0,4 UI of oxytocin until obstetrician determines that uterine tone is adequate.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Intravenous bolus infusion of oxytocin 3UI followed by re-asessment of uterine tone by obstetrician after 3 minutes. Infusion stops when uterine tone is adequate and is repeated if inadequate to the maximum of 9UI (3 bolus infusions). If uretine tone is inadequate after 9UI then other methods for preventing bleeding will be used.

SUMMARY:
Introduction: postpartum hemorrage is a leading cause of death after cesarean sections in Brazil. Oxytocin is the main drug for both prophylaxis and threatment of postpartum hemorrage because uterine atony is the most prevalent cause. Both excessive and too low oxytocin doses threaten the life of women.

Objective: to determine the minimum effective dose of oxytocin for cesareans during labor.

Method: adaptative clinical trial using a modified up and down method of two sequential groups: rule of three and continuous infusion. Allocation in rule of three or continuous infusion will be random and masked for patients and anesthesiologists. The minimum effective dose will be the effective dose for 90% of success (ED90 for preventing uterine atony).

ELIGIBILITY:
Inclusion Criteria:

* Cesarean delivery during labor.
* Spinal anesthesia

Exclusion Criteria:

* Change of anesthesia

Ages: 18 Years to 130 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Oxytocin dose | 10 minutes
  Minumum oxytocin dose for preventing uterine atony in 90% of cesareans.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário de Brasília, Brasília, Federal District, Brazil